CLINICAL TRIAL: NCT05491408
Title: Effect of Cough Assist Device in COPD Patients Admitted to Respiratory Intensive Care Unit at Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebtesam Adel Hammad Askar, principal investigator, Assiut University
Other Study IDs: cough assist device in ICU
Record Dates: First submitted 2022-07-22; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients exposed to cough assist device: the first group will include patients with COPD who received conventional management in addition to cough assist device
  Interventions: Device: Cough assist device
- patients not exposed to cough assist device: the second group will include COPD patients who received conventional management only.

INTERVENTIONS:
Device: Cough assist device — A device that facilitates airway secretion clearance in COPD patients, thus avoiding hospitalisations and preventing pneumonias and episodes of respiratory failure [4,5].
  Groups: patients exposed to cough assist device

SUMMARY:
1. To evaluate the effecacy of cough assist device (CAD) in COPD patients admitted in RICU either on invasive or Non-invasive ventilation.
2. To detect any possible complications associated with the use of cough assist device.

DETAILED DESCRIPTION:
Effective cough is a protective mechanism against respiratory tract infections. COPD patients may have impaired cough and a reduction in peak cough flows(PCF) as a result of inspiratory and expiratory muscle weakness, which causes a reduction in the pressure available to drive the cough manoeuver.

Cough augmentation with mechanical Insufflation-Exsufflation (MI-E) has been described as a technique that facilitates airway secretion clearance in COPD patients, thus avoiding hospitalisations and preventing pneumonias and episodes of respiratory failure .

Cough augmentation techniques comprise lung volume recruitment, (also termed air stacking or breaths tacking), mechanically assisted cough using mechanical insufflation-exsufflation (MI-E) device. During lung volume recruitment, the person inhales a volume of gas via the ventilator, or self-inflating resuscitation bag adapted with a one-way valve to facilitate gas holding. The person retains the inhaled volume by closing the glottis, inhales another volume of gas and then again closes the glottis; this process is repeated until maximum insufflation capacity is reached MI-E devices deliver a positive (inflation) and negative pressure (rapid deflation) delivered to the person via an oronasal interface, mouthpiece, or endotracheal or tracheostomy tube. MI-E comprises a pressure -targeted lung insufflation followed by vacuum exsufflation, enabling lung emptying and increasing peak cough flow. Alternation of pressure may be manually or automatically cycled. Pressures of 40 mmHg (insufflation) to 40 mmHg (exsufflation) (54 cmH2O) are usually most effective and best tolerated by the person .

Treatments usually comprise three to five insufflation-exsuflation cycles followed by a short period of rest to avoid hyperventilation. Treatments can be repeated until no further secretions are expectorated. MIE can be performed in isolation or in combination with manually assisted cough .

Few complications associated with MI-E devices as a drop in oxygen levels, barotrauma elevated blood pressure for more than 30 minutes have been reported, most likely due to use of pressures that are much lower than physiological cough pressures and the short duration of application .

ELIGIBILITY:
Inclusion Criteria:

* All COPD patients above 18 years old who admitted to RICU.

Exclusion Criteria:

* • All patients who have: neuromuscular diseases, pulmonary oedema, cardiac arrest, cardiogenic shock, acute myocardial infarction, pneumothorax, pulmonary neoplasm, pulmonary thromboembolism.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All Patient Will be subjected to:
  1. Detailed clinical history &physical examination.
  2. Hemodynamics assessment.
  3. GCS assessment.
  4. Routine investigations.
  5. Using Cough Assisted device in the first group: Settings of the Cough Assist device (inhale, exhale pressure, insufflation time, inhale flow).
  6. Clinical assessment of patients before and after use of CAD including : RR, intensity of rhonchi and crepitations accessory muscle use,asynchrony with the machine either invasive or non-invasive.
  7. ABG before and after use CAD
  8. Physiological assessment of the patient including PEEP, plateau pressure, resistance and compliance before and after application of CAD in mechanically ventilated patients.
  9. Calculation the amount of secretion before and after using CAD.
  10. The duration of MV and the length of RICU stay will recorded.
  11. Any possible complications will be recorded including drop in oxygen levels, barotrauma elevated blood pressure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of Cough Assist Device (CAD) in COPD patients admitted in RICU including need for invasive or Non-invasive ventilation and weaning success. | Baseline
  number of COPD patients who are on NIV that no further in need for MV after use of cough assist device will be calculated also number of COPD patients who are on MV , we will assess early weaning , rate of mortality among them after use of cough assist device in this group of patients